CLINICAL TRIAL: NCT00735553
Title: A Phase III, Three-arm, Parallel Design, Placebo-controlled, Randomized, Double-blind, Multicenter Study Evaluating the Safety and Efficacy of Proellex® (CDB-4124) in the Treatment of Premenopausal Women With Symptomatic Uterine Fibroids
Brief Title: Evaluating the Safety and Efficacy of Proellex® (CDB-4124) in Premenopausal Women With Symptomatic Uterine Fibroids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Repros stopped the study for safety and FDA put the study on hold for safety.
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZPU-303
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Uterine Fibroids
Keywords: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 25 mg Proellex (Active Comparator): 25 mg oral daily dose of Proellex
  Interventions: Drug: Proellex
- 50 mg Proellex (Active Comparator): 50 mg oral daily dose of Proellex
  Interventions: Drug: Proellex
- placebo (Placebo Comparator): oral daily dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proellex — One 25 mg capsule of Proellex® and one placebo capsule orally daily for up to four months
  Other Names: Telapristone acetate
  Arms: 25 mg Proellex
Drug: Proellex — Two 25 mg mg capsules of Proellex® orally daily for up to four months
  Other Names: Telapristone acetate
  Arms: 50 mg Proellex
Drug: Placebo — Two placebo capsules orally daily for up to four months
  Other Names: Sugar pill
  Arms: placebo

SUMMARY:
Premenopausal women with symptomatic uterine fibroids will be randomized to either Proellex 25mg or 50mg or placebo for one treatment cycle (four months). Safety and effectiveness between 50 mg versus placebo, and between 25mg and placebo will be analyzed.

DETAILED DESCRIPTION:
Subjects with documented uterine fibroids, screening UFS-QOL severity score of at least 40, and meeting other eligibility criteria will be enrolled in the study. Following screening and a pre-treatment endometrial biopsy, subjects will be assessed monthly for the four (4) month double-blinded treatment phase. The study duration is approximately six months, comprised of a one-month screening period, 4 month treatment period and one month follow-up period. Subjects' blood will be drawn in a fasting state to obtain the pre-dose trough (PK) levels of study drug at each study drug dosing/dispensation visit to determine the potential for drug accumulation.

ELIGIBILITY:
Inclusion Criteria:

* Speak, read and understand English or Spanish;
* Not have undergone hysterectomy, uterine arterial embolization or endometrial ablation therapy (previous myomectomy is acceptable) for any cause and no surgical interventions for uterine fibroids (e.g. hysterectomy, myomectomy, uterine arterial embolization) are planned or anticipated during the study;
* One uterine fibroid must be identifiable and measurable by transvaginal ultrasound;
* Menstrual cycle lasting from 24 to 36 days;
* History of excessive menstrual bleeding;
* Negative urine pregnancy test at screening.

Exclusion Criteria:

* Six months or more (immediately prior to Screening Visit) without a menstrual period;
* Prior hysterectomy;
* Prior bilateral oophorectomy;
* Pregnant or lactating females or women who are attempting or expecting to become pregnant at any time during the study;
* Documented endometriosis, active pelvic inflammatory disease (PID), platelet dysfunction, or Von Willebrand's Disease;
* Any history or diagnosis of gynecological cancer or cervical dysplasia of any grade including atypical squamous cells of undetermined significance (ASCUS) associated with Human Papilloma Virus (HPV);
* Subject with diagnosed or suspected carcinoma of the breast, reproductive organs or any other organ system;
* Subject with known active infection with HIV, Hepatitis A, B or C, Gonorrhea, or Chlamydia or previous history of auto-immune disease or positive serum antinuclear antibodies.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andre vanAs, MD, PhD, Study Director — Repros Therapeutics Inc.
Locations (15):
- United States (15):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Women's Health Care at Frost Steet, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - OB-GYN Associates of Mid-Florida, P.A., Leesburg, Florida
  - Miami Research Associates, Miami, Florida
  - Insignia Clinical Research, Tampa, Florida
  - SC Clinical Research Center, Columbia, South Carolina
  - Advanced Research Associates, Corpus Christi, Texas
  - Advances in Health Inc., Houston, Texas
  - The Woman's Hospital of Texas, Clinical Research Center, Houston, Texas
  - Institute for Women's Health, San Antonio, Texas
  - Seven Oaks Women's Ctr., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- All Groups: 25 mg, 50 mg oral daily dose of Proellex or placebo
Period: Overall Study
Arm/Group | All Groups
Started | 77
Completed | 0
Not Completed | 77
Not completed — Study prematurely terminated | 77

BASELINE CHARACTERISTICS:
Population: Study prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg Proellex | 50 mg Proellex | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Efficacy of 50 mg Proellex® Versus Placebo in the Treatment of Subjects With Symptomatic Uterine Fibroids From Baseline to Month 4 as Determined by Scoring Changes in the Pictorial Blood Loss Assessment Chart (PBAC)
Time Frame: 4 months
Population: Study prematurely terminated
Arm/Group | 25 mg Proellex | 50 mg Proellex | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: No adverse event data is available.
Arm/Group | 25 mg Proellex | 50 mg Proellex | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated for safety reasons (Proellex studies were put on clinical hold due to liver toxicity). Sponsor was unable to pay vendor, and was therefore not provided with any study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights